CLINICAL TRIAL: NCT04388410
Title: Phase 2b/3 Trial to Evaluate the Safety and Efficacy of Plasma Transfusion From Convalescent Patients With SARS-CoV-2 Infection on Severity and Mortality of COVID-19 in Hospitalized Patients.
Brief Title: Safety and Efficacy of Convalescent Plasma Transfusion for Patients With COVID-19
Acronym: EPCOvid-1
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: TecSalud Investigación Clínica (Other); Instituto Nacional de Enfermedades Respiratorias (Other Government); Instituto Nacional de Cardiologia Ignacio Chavez (Other); Hospital General Dr. Manuel Gea González (Other Government); Hospital Regional de Alta Especialidad del Bajio (Other); Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Juan G. Sierra Madero, Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3380
Record Dates: First submitted 2020-05-12; First posted 2020-05-14 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; convalescent plasma; randomized clinical trial
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, multicenter, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Encasement of plasma and saline bags with an identical material will be done in Blood bank
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- convalescent plasma (Experimental): Convalescent plasma obtained from volunteers who have recovered from COVID 19. Enclosed with a similar material as the control
  Interventions: Biological: convalescent plasma
- Normal saline (Placebo Comparator): Normal saline solution in 200 ml plasma bags enclosed with with a similar material as the plasma
  Interventions: Biological: convalescent plasma

INTERVENTIONS:
Biological: convalescent plasma — Plasma obtained from volunteers who have recovered from SARS-Cov-2 infection. Two 200 ml infusions will be administered with 24-72 hours in between.

SUMMARY:
This is a multicenter double blinded study to evaluate the efficacy and safety of convalescent plasma from COVID-19 recovered individuals to treat hospitalized patients with severe COVID-19 disease. The study will enroll 410 subjects who will be randomized 1:1 to receive convalescent plasma or normal saline solution in a blinded manner. The primary endpoint will be improvement on the 8 point WHO scale over 28 days. Mortality at day 28 will be a secondary endpoint. An interim analysis will be done when 224 patients have completed their follow up to assess safety and to indicate continuation or stopping of the study, based on safety and efficacy observed.

DETAILED DESCRIPTION:
A total of 410 patients with COVID 19 who fulfill inclusion criteria will be invited to receive:

Human convalescent plasma from recovered patients in two infusions of 200 ml separated with 24 to 72 hours or Normal saline solution in a similar plasma bag. Both products will be covered in an identical material to avoid identification of the infused product.

Primary endpoint:

Improvement on the 8 point WHO scale over 28 days.

Secondary endpoints.

Mortality at day 28

* Presence of antibodies against SARS-CoV-2 in serum on days 0, 3, 7, 14, 21 y 28 after plasma administration, as long as the patient remains in the hospital.
* Disease progression to a worse stage compared to the baseline on admission to the study according to SOFA scale.
* Disease progression to a worse stage defined as worsening in at least two categories in the OMS disease scale on different timelines in comparison to baseline on admission to the study
* Number of hours on mechanical ventilation in those who enter the study on mechanical ventilation.
* Number of days with fever defined as temperature >38°C on at least one occasion during the day

Inclusion criteria:

1. Adults older than 18 years.
2. Confirmed SARS-CoV2 infection
3. Patient hospitalized for COVID 19
4. Severe disease or risk for severe disease
5. Informed consent from patient or responsible person.

Exclusion criteria

1. History of allergic reactions to blood products
2. SOFA scale >12 points
3. Absolute contraindication for administration of plasma
4. Participation in other blinded clinical trial
5. Projected life expectancy less than 3 months
6. Any condition perceived by the investigator as not appropriate for participation of the patient in the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years of age and older.
2. Confirmed SARS-CoV2 infection
3. Hospitalized for COVID 19
4. Severe disease or risk for severe disease
5. Informed consent from patient or responsible person.

Exclusion Criteria:

1. History of allergic reactions to blood products
2. SOFA scale >12 points
3. Absolute contraindication for administration of plasma
4. Participation in other blinded clinical trial
5. Projected life expectancy less than 3 months
6. Any condition perceived by the investigator as not appropriate for participation of the patient in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Severity and death | 28 days
  Ordinal 8-point severity outcome scale: 1 Death, 2 Hospitalized, intubated and receiving mechanical ventilation and additional organ support (eg. renal replacement therapy, vasopressors, extracorporeal membrane oxygenation), 3 Hospitalized, intubated and receiving mechanical ventilation but no additional organ support, 4 Hospitalized receiving non-invasive ventilation of high-flow oxygen, 5 Hospitalized, receiving supplementary oxygen by mask or nasal prongs, 6 Hospitalized, no oxygen therapy needed, 7 Not-hospitalized (ambulatory) with limited activity, 8 Not-hospitalized (ambulatory) with no limitation of activities.
Adverse events that require study treatment interruption | During the 28 day of follow up
  Any unfavorable and unintended symptom or sign (including an abnormal laboratory finding) temporally associated with the study intervention and considered related to the intervention that require interruption of study treatment. Including but not limited to: Severe allergic reactions (rash and fever), transfusion-associated lung injury (TRALI), transfusion-associated circulatory overload (TACO), and other severe unexpected events

SECONDARY OUTCOMES:
Time to clinical improvement | 28 days
  Time (in days) to improvement in at least two categories in the 8-point ordinal severity scale in comparison to baseline on admission to the study.
Severity and death | Days 1, 3, 5, 7, 12, 14, and 21.
  Ordinal 8-point severity outcome scale: 1 Death, 2 Hospitalized, intubated and receiving mechanical ventilation and additional organ support (eg. renal replacement therapy, vasopressors, extracorporeal membrane oxygenation), 3 Hospitalized, intubated and receiving mechanical ventilation but no additional organ support, 4 Hospitalized receiving non-invasive ventilation of high-flow oxygen, 5 Hospitalized, receiving supplementary oxygen by mask or nasal prongs, 6 Hospitalized, no oxygen therapy needed, 7 Not-hospitalized (ambulatory) with limited activity, 8 Not-hospitalized (ambulatory) with no limitation of activities.
Antibodies against SARS-CoV-2 | Days 0, 3, 7, 14, 21, 28
  Antibody titers on serum/plasma as long as the patient remains in the hospital.
Disease progression 1 | 28 days
  Changes in SOFA scale during hospitalization compared to the baseline
Disease progression 2 | Days 7,14, 21, 28
  Changes in at least two categories in the 8-point ordinal severity scale in comparison to baseline on admission to the study
Time on mechanical ventilation | 28 days
  Time (in hours) spent receiving invasive mechanical ventilation in those who enter the study on mechanical ventilation.
Number of days with fever | 28 days
  Temperature >=38°C on at least one measurement during the day
Adverse events attributed to the study intervention | 28 days
  Any unfavorable and unintended symptom or sign (including an abnormal laboratory finding) temporally associated with the study intervention and considered related to the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Juan G Sierra-Madero, MD, Principal Investigator — Department of Infectious Diseases
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No
Plan to make IPD still not decided and would need approval by regulatory authorities